CLINICAL TRIAL: NCT01095172
Title: A Randomized Trial of Rituximab in Induction Therapy for Living Donor Renal Transplantation
Brief Title: RituxiMab INDuction in Renal Transplantation
Acronym: ReMIND
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Principal Investigator, Nizam Mamode, Consultant Surgeon and Reader in Transplant Surgery, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RituxiRT; 2009-017066-23 (EudraCT Number); 95769119 (Registry Identifier: ISRCTN); 9154 (Registry Identifier: UK Clinical Research Network (CRN) Portfolio)
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Function of Renal Transplant
Keywords: Immunosuppression; Rituximab; B cell
MeSH Terms: interventions — Rituximab; Tacrolimus; Mycophenolic Acid; Hydrocortisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Rituximab 375mg/m2
  Low dose tacrolimus with mycophenylate mofetil, hydrocortisone and 1 week prednisolone
  Interventions: Drug: Rituximab; Drug: Tacrolimus; Drug: Mycophenylate mofetil; Drug: Hydrocortisone; Drug: Prednisolone
- Control group (Active Comparator): Low dose tacrolimus with mycophenylate mofetil and continued prednisolone
  Interventions: Drug: Tacrolimus; Drug: Mycophenylate mofetil; Drug: Hydrocortisone; Drug: Prednisolone

INTERVENTIONS:
Drug: Rituximab — 375mg/m^2, single dose given 2-4 weeks prior to transplantation
  Other Names: Mabthera
  Arms: Rituximab
Drug: Tacrolimus — dose calculated to give levels of 3-7ng/ml
  Other Names: Advagraf, Adoport, Prograf
Drug: Mycophenylate mofetil — Mycophenylate mofetil 2g/day in divided doses
  Other Names: MMF, Cellcept
Drug: Hydrocortisone — 100mg hydrocortisone on the evening of the day of surgery and 2 further doses of hydrocortisone on day 1 post transplant.
Drug: Prednisolone — Prednisolone 0.3mg/kg on day 2, 0.25mg/kg on day 3, 0.2mg/kg on day 4 and 0.16mg/kg on day 5. On day 6 they will receive 5mg prednisolone, and on day 7 none.
  Arms: Rituximab
Drug: Prednisolone — Reducing dose of prednisolone over at least 6 months. Subsequent steroid maintenance or withdrawal will be at the discretion of the patient's clinician.
  Arms: Control group

SUMMARY:
Hypothesis:

* That B cell depletion, rather than reducing acute rejection, will allow minimisation of immunosuppression, which may lead to better graft survival.

Aim:

* To assess whether the addition of rituximab to a low-dose tacrolimus immunosuppression regime allows a reduction in steroid administration.

Objectives:

* To assess whether B cell depletion affects graft function, acute rejection and complication rates
* To assess whether the T cell response to allotransplantation is impaired by B cell depletion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years receiving their first living donor renal transplant, or their second if the first was not lost from acute rejection
* Patients who have given written informed consent
* Women of child bearing potential taking adequate contraception.

Exclusion Criteria:

* Previous other organ transplants lost through acute rejection
* Patients undergoing antibody incompatible transplantation
* Patients with other organ transplants
* Patients previously treated with cyclophosphamide, ATG, OKT3 or rituximab
* Patients with white cell count below 4.0x10^9/L.
* Patients with platelet count below 100x10^9/L
* Patients who are treated with drugs that are strong inhibitors or inducers of cytochrome P450, or treated with terfenadine, astemizole, cisapride or lovastatin
* Patients who have been involved in any other investigational trial or non protocol immunosuppressive regimen in the previous 90 days prior to transplant
* Pregnant or breastfeeding women
* Patients with a documented history of malignancy and its origins and treatment in the last five years. (Localised basal cell carcinoma of the skin is permitted)
* Patients known to be HIV, Hepatitis B surface antigen or Hepatitis C antibody positive
* Patients who in the opinion of the Investigator would not be a suitable candidate for study participation
* Women of child bearing potential not willing to take adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2020-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Estimated GFR (calculated using the Cockcroft-Gault formula) | 1 year

SECONDARY OUTCOMES:
Biopsy proven acute rejection (based on Banff classification) | 1, 2, 3, 4, 5 years
Allograft survival | 1, 2, 3, 4, 5 years
Patient Survival | 1, 2, 3, 4, 5 years
Infection rate | 1 year
  New episodes, including (but not restricted to) viral (e.g. CMV, EBV), bacterial (e.g. Urinary Tract Infections with details of causative organism) and fungal infections will be recorded at each assessment time-point.
Changes in B and T cell repertoire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nizam Mamode, MD FRCS(Gen), Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - South West Transplant Centre, Plymouth, Devon
  - East Kent Hospitals NHS Foundation Trust, Canterbury, Kent
  - Glasgow Renal and Transplant Unit, Glasgow
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Sheffield Kidney Institute, Sheffield